CLINICAL TRIAL: NCT06474325
Title: Feasibility and Acceptability of Mobile Mental Health Application for the Improvement of Medication Adherence in Persons With Schizophrenia(SZ) and Schizoaffective Disorder(SZA)
Brief Title: Feasibility and Acceptability of Mobile Mental Health App for SZ and SZA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Government Medical College, Palakkad-678013 (Unknown)
Responsible Party: Principal Investigator, Vishwajit Nimgaonkar, MD PhD, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY23090042; D43TW009114 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Schizo Affective Disorder
Keywords: Schizophrenia; Schizo Affective Disorder; Adherence; Mobile app
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: To compare the Medication adherence rating scale scores before and after using mental health application for improving medication adherence in persons with schizophrenia and schizoaffective disorder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention via mobile app (Experimental): Intervention via mobile application include psychoeducational videos, reminders, and virtual rewards and badges for completing the challenges to encourage adherence of medications
  Interventions: Behavioral: Intervention via mobile application

INTERVENTIONS:
Behavioral: Intervention via mobile application — Intervention via mobile application include psychoeducational videos, reminders, and virtual rewards and badges for completing the challenges to encourage adherence of medications

SUMMARY:
A new mental health application will be developed for persons with schizophrenia and schizoaffective disorder. The aim is to look at whether it is feasible to use a mobile health application for improving medication adherence in persons with schizophrenia and schizoaffective disorder and whether it is acceptable to that population.

DETAILED DESCRIPTION:
Many interventions have been tried to improve the medication adherence of patients with schizophrenia. Individualized interventions using like setting alarms and using checklists have shown significant improvement in compliance with the medications. In the era of mobile applications most of the persons use mobile applications for multiple purposes, which have the potential to influence the life of a person in many ways. A meta-analysis conducted in 2016 showed that 66.4% of psychotic patients owned a mobile phone. A study conducted in North India found that 84.4% of patients with severe mental disorders owned a mobile phone. So if used properly it can also help in improving the life of a person with SZ.

Many mobile applications have been used to improve medication compliance in general. But only a few mobile applications have specifically focused the persons with schizophrenia. Very few studies have investigated the efficacy of mobile applications to improve medication adherence in patients with schizophrenia. This study will be assessing the feasibility of developing a mobile application and using the application for improving compliance of medications in persons with schizophrenia and schizoaffective disorder.

Primary aims:

* To develop a mobile mental health application for the improvement of medication adherence in persons with schizophrenia and schizoaffective disorder
* To assess the feasibility and the acceptability of using a mobile mental health application for improving the medication adherence of persons with schizophrenia and schizoaffective disorder

Primary Objectives:

• To assess the feasibility and the acceptability of using a mobile mental health application for improving the medication adherence of persons with schizophrenia and schizoaffective disorder

Secondary Objective:

• To compare the Medication adherence rating scale scores before and after using mental health application for improving medication adherence in persons with schizophrenia and schizoaffective disorder

1. Initial screening of the participants will be done by the psychiatrist( PI)( In the Psychiatry OPD )
2. Persons with schizophrenia and schizoaffective disorder who are in remission(In Remission for past 2 months) and attending the Psychiatry Outpatient department at Government Medical College, Palakkad will be recruited
3. After taking informed consent participants will be assigned into intervention group
4. Pre intervention assessments will be done ((e.g., Symptoms, the Medication Adherence using relevant scales)
5. After the pre-intervention assessment, Mobile application will be installed into participants mobile phone(Instruction will be given on the features of the mobile application and how to use it )
6. Participants will receive the intervention via mobile application installed to their mobile phone (patient will continue to take their regular medications including antipsychotics. Intervention via mobile application include psychoeducational videos, reminders, and virtual rewards and badges for completing the challenges to encourage adherence of medications)
7. Duration of intervention will be three months
8. Post-intervention assessment will be done within one week after completion of the intervention (e.g., symptoms, the Medication Adherence, feedback (Acceptance questionnaire)

ELIGIBILITY:
Inclusion Criteria:

1. Persons diagnosed with schizophrenia and schizoaffective disorder and are in remission for past two months.
2. Age 18-60 years of any gender.
3. Able to read and understand Malayalam/ English

Exclusion Criteria:

1. Patients who have active psychotic or mood symptoms.
2. History of substance use (except nicotine)
3. Having any serious physical illness. -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Mobile app | Baseline and after three months
  To assess the feasibility and the acceptability with a mobile mental health application for medication adherence in persons with SZ and schizoaffective disorder using Acceptability Questionnaire. The scale ranges from 0 to 50.
Acceptibility of Mobile app | Baseline and after three months
  To assess the feasibility and the acceptability with a mobile mental health application for medication adherence in persons with SZ and schizoaffective disorder using Perception of treatment Acceptability scale (Score (0-5) 0= Not at all 5 =very much). Ranges from 0 to 50.
  )
Adherence to medication | Baseline and after three months
  To compare the Medication adherence rating scale scores before and after using mental health application for changing medication adherence in persons with schizophrenia and schizoaffective disorder

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit Nimgaonkar, MD, PhD, Principal Investigator — University of Pittburgh
Locations (1):
- Government Medical College,, Palakkad, Kerala, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: One year after publication of this study.
Access Criteria: For individual participant data, meta-analysis.